CLINICAL TRIAL: NCT00039273
Title: An Open Label Phase II Clinical Trial To Evaluate The Safety And Efficacy Of ABX-EGF In Patients With Metastatic Colorectal Carcinoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069368; UCLA-0112063; IMMUNEX-054-0005; NCI-G02-2073
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab

INTERVENTIONS:
Biological: panitumumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have relapsed or refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with metastatic colorectal cancer treated with monoclonal antibody ABX-EGF.
* Determine the additional measures of clinical efficacy of this drug, in terms of progression-free survival, overall survival, and time to treatment failure, in these patients.
* Determine the safety of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive monoclonal antibody ABX-EGF IV over 1 hour weekly on weeks 1-8. Treatment repeats every 8 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, every 3 months for 1 year, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 20-100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal carcinoma

  * Diagnosed by fine-needle aspirate or tissue biopsy
  * Metastatic disease
  * No squamous cell carcinoma
* Relapsed or refractory after prior chemotherapy with irinotecan and a fluoropyrimidine (i.e., fluorouracil, capecitabine, or ftorafur with or without leucovorin calcium) given concurrently or sequentially

  * Progressive disease within 2 months of last dose of this prior chemotherapy for metastatic disease OR
  * Evidence of relapse within 12 months after last dose of adjuvant therapy
* Bidimensionally measurable disease
* Overexpression of epidermal growth factor r (EGFr) by immunohistochemistry

  * Must be 2+ or 3+ in at least 10% of evaluated tumor cells
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.2 mg/dL

Cardiovascular:

* LVEF at least 45% by MUGA
* No myocardial infarction within the past year

Other:

* HIV negative
* No other malignancy within the past 5 years except basal cell carcinoma or carcinoma in situ of the cervix
* No chronic medical or psychiatric condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior EGFr-targeting agents or biological agents with antitumor activity

Chemotherapy:

* See Disease Characteristics
* At least 30 days since prior systemic chemotherapy
* No more than 2 prior fluoropyrimidine regimens (e.g., fluorouracil and leucovorin calcium followed by capecitabine)
* No other prior chemotherapy, except leucovorin calcium, for colorectal carcinoma

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 30 days since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 30 days since other prior anticancer therapy
* No prior investigational drug with potential antitumor activity
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-07; Primary Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Randolph Hecht, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Meropol NJ, Berlin J, Hecht JR, et al.: Multicenter study of ABX-EGF monotherapy in patients with metastatic colorectal cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1026, 256, 2003.